CLINICAL TRIAL: NCT02877784
Title: Determination of Accurate Screening Tools for Dysphagia in Oculopharyngeal Muscular Dystrophy
Brief Title: Screening in Oculopharyngeal Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601374
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Oculopharyngeal Muscular Dystrophy
Keywords: screening; OPMD; dysphagia; dysarthria
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal; Deglutition Disorders; Dysarthria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening: Participants enrolled will undergo testing of the swallowing mechanism
  Interventions: Procedure: Videofluoroscopic swallowing study; Other: Functional Oral Intake Scale; Other: Eating Assessment Tool-10

INTERVENTIONS:
Procedure: Videofluoroscopic swallowing study — Videofluoroscopic swallowing study will be performed to measure the oropharyngeal swallowing.
  Other Names: VFSS; modified barium swallow (MBS)
Other: Functional Oral Intake Scale — The Functional Oral Intake Scale (FOIS) will be used for participants to report their food intake habits.
  Other Names: FOIS
Other: Eating Assessment Tool-10 — The Eating Assessment Tool-10 will be used for participant reporting of swallowing system severity.
  Other Names: EAT-10

SUMMARY:
Oculopharyngeal muscular dystrophy (OPMD) is a rare myopathic disease that results in progressive degeneration of the oral and pharyngeal muscular, resulting in severe dysphagia and dysarthria. OPMD is considered a rare disease; therefore, limited research is available on the natural progression of the disease or the utility of biomarkers to identify swallowing impairment. The aim of this study is:

1. To identify accurate, reliable and non-invasive clinical markers of swallowing impairment
2. To determine the discriminate ability of these markers to identify impairments in swallow safety and swallowing efficiency.

DETAILED DESCRIPTION:
Participants will be recruited from the Neurology clinic at the University of Florida. The single evaluation will occur in the PIs research laboratory at the University of Florida, Gainesville, Florida.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of oculopharyngeal muscular dystrophy
* no allergies to barium or capsaicin,
* no tracheotomy or mechanical ventilation
* no significant concurrent respiratory disease (e.g., COPD).

Exclusion Criteria:

* Pregnant Women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample population will consist of individuals with a diagnosis of oculopharyngeal muscular dystrophy.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Dynamic Imaging Grade of Swallowing Toxicity | Baseline
  Global Metric of swallowing Safety and Efficiency

SECONDARY OUTCOMES:
Dietary intake as confirmed by Functional Oral Intake Scale (FOIS) | Baseline
  FOIS is a validated 7-point scale indexing an individual's ability to intake food on a day-to-day basis.
  TUBE DEPENDENT (levels 1-3) No oral intake Tube dependent with minimal/inconsistent oral intake Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7) Total oral intake of a single consistency Total oral intake of multiple consistencies requiring special preparation Total oral intake with no special preparation, but must avoid specific foods or liquid items Total oral intake with no restrictions
Participant perception of swallowing related symptoms as confirmed by The Eating Assessment Tool 10 (EAT-10) | Baseline
  EAT-10 is a 10-item validated self-administered dysphagia severity symptom survey. Score is 0 - 40 with 0 being the best possible score and 40 the worst possible score.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States